CLINICAL TRIAL: NCT04004793
Title: Effect of Dapagliflozin for Remission of Type 2 Diabetes Mellitus: A Multicenter, Randomized, Placebo-Controlled Trial
Brief Title: Remission of Type 2 Diabetes With Dapagliflozin (READ Trial)
Acronym: READ
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Xiaoying Li, Professor, Medical doctor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZSE-201901
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin plus intensive lifestyle intervention (Experimental): The treatment of Dapagliflozin (Forxiga®) will be initiated and maintained at 10mg every morning until the completion of the study.
  Interventions: Behavioral: Intensive lifestyle intervention; Drug: Dapagliflozin 10 MG Oral Tablet
- Placebo plus intensive lifestyle intervention (Placebo Comparator): The treatment of placebo will be initiated and maintained at 10mg every morning until the completion of the study.
  Interventions: Behavioral: Intensive lifestyle intervention; Drug: Placebo Oral Tablet

INTERVENTIONS:
Behavioral: Intensive lifestyle intervention — Participants were will be asked to follow a weight management programme, in accordance with the American Diabetes Association guidelines. Weight loss will be induced with a diet replacement phase using an energy restriction diet (energy deficit by 500~750 kcal/day) for 3 months, with <35% as fat, >15% as protein. The minimum energy intake is 1200kcal/day for men and 1000kcal/day for women.. Additionally, participants were encouraged to increase physical exercise (≥150 minutes of brisk walking every week or ≥10000 steps per day).
Drug: Dapagliflozin 10 MG Oral Tablet — The treatment of Dapagliflozin (Forxiga®) will be initiated and maintained at 10mg every morning until the completion of the study.
  Arms: Dapagliflozin plus intensive lifestyle intervention
Drug: Placebo Oral Tablet — The treatment of placebo will be initiated and maintained at 10mg every morning until the completion of the study.
  Arms: Placebo plus intensive lifestyle intervention

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study to assess the effect of dapagliflozin add-on intensive lifestyle intervention for remission of type 2 diabetes in obese patients with Type 2 Diabetes Mellitus. The study consists of a 12-months treatment period (in which they will receive either Dapagliflozin plus intensive lifestyle intervention or placebo plus intensive lifestyle intervention in addition to the background therapy), and a 2-month follow-up period after treatment period.

DETAILED DESCRIPTION:
Diabetes remission is an important issue which has not been well studied. Some studies showed that bariatric surgery and intensive lifestyle intervention could lead to remission in diabetic patients. Our present study aims to assess the effect of dapagliflozin add-on intensive lifestyle intervention on remission of type 2 diabetes in obese patients with type 2 diabetes. This is a multicenter, randomized, double-blind, placebo-controlled study. The study consists of a 12-months treatment period (in which subjects will receive either dapagliflozin plus intensive lifestyle intervention or placebo plus intensive lifestyle intervention in addition to the background therapy), and a 2-month follow-up period after treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 20-70 years old who had a BMI ≥25 kg/m2.
* Subjects had been diagnosed with type 2 diabetes within 6 years
* HbA1C ≥6.5% and ≤10.0% at screening if on treatment with metformin alone or without antidiabetic agents, or HbA1C <6.5% at screening if on metformin treatment alone
* Able and willing to provide written informed consent and to comply with the study

Exclusion Criteria:

1. Patients have a history of myocardial infarction, unstable angina, cardiac surgery or revascularization (coronary artery bypass graft/percutaneous transluminal coronary angioplasty), or congestive heart failure New York Heart Association Class III or IV.
2. Current insulin use.
3. Weight loss of more than 5kg within the past 6 months.
4. Women who are pregnant or plan to become pregnant.
5. Diagnosis or history of acute metabolic diabetic complications such as ketoacidosis or hyperglycemic hyperosmolar state, or diabetes insipidus within 30 days.
6. Alcohol or drug abuse within the 3 months prior to informed consent that would interfere with trial participation or any ongoing condition leading to a decreased compliance to study procedures or study drug intake.
7. Intake of an investigational drug in another trial within 30 days prior to intake of study medication in this trial or participating in another trial (involving an investigational drug and /or follow-up).
8. Patients with clinically apparent hepatobiliary disease, including but not limited to chronic active hepatitis and/or severe hepatic insufficiency. ALT or AST > 3x upper limit of normal (ULN), or serum total bilirubin (TB) >34.2 μmol/L (>2 mg/dL).
9. Patients with severe renal impairment or end-stage renal disease (eGFR< 45 mL/min/1.73 m2).
10. Bariatric surgery within the past two years and other gastrointestinal surgeries that induce chronic malabsorption.
11. Malignancy within 5 years of the enrollment visit.
12. Known immunocompromised status, including but not limited to, individuals who had undergone organ transplantation or acquired immunodeficiency syndrome (AIDS).
13. History of bone fracture secondary to diagnosed severe osteoporosis.
14. Current treatment with systemic steroids at time of informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent or any other uncontrolled endocrine disorder except T2DM.
15. Administration of sibutramine, phentermine, orlistat, rimonabant, benzphetamine, diethylpropion, methamphetamine, or phendimetrazine within 30 days of enrollment visit.
16. Blood dyscrasias or any disorders causing haemolysis or unstable Red Blood Cell (e.g. malaria, babesiosis, haemolytic anaemia).
17. Administration of any other investigational drug within 30 days of planned enrollment to this study, or within 5 half-life periods of other investigational drugs.
18. Subject is, in the judgment of the Investigator, unlikely to comply with the protocol or has any severe concurrent medical or psychological condition that may affect the interpretation of efficacy or safety data

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of patients with diabetes remission | During the 12-month intervention
  Diabetes remission is defined as a HbA1c<6.5% and a fasting glucose level of <7.0 mmol/l in the absence of all antidiabetic medication for at least 2 months

SECONDARY OUTCOMES:
Proportion of patients with diabetes remission | during the 12-month intervention
Net change in body weight | during both 12 and 14 months
Net change in waist circumference | during both 12 and 14 months
Net change in HOMA-IR | during both 12 and 14 months
Net change in serum lipids | during both 12 and 14 months
Net change in HbA1c | during both 12 and 14 months
Net change in body fat | during both 12 and 14 months
Net change in SBP | during both 12 and 14 months
Net change in Serum Creatine | during both 12 and 14 months
Net change in Albuminuria | during both 12 and 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, MD, Principal Investigator — Fudan University
Locations (1):
- Shanghai Medical college of, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Y, Chen Y, Ma J, Lin J, Liu C, Li X, Xu Y, Kuang H, Shi L, Xue Y, Feng B, Zhu D, Wang G, Yang J, Xiao X, Yu X, Zhou J, Bao Y, Su Q, Lyu M, Li X, Zhang H, Li X. Dapagliflozin plus calorie restriction for remission of type 2 diabetes: multicentre, double blind, randomised, placebo controlled trial. BMJ. 2025 Jan 22;388:e081820. doi: 10.1136/bmj-2024-081820. PMID 39843169